CLINICAL TRIAL: NCT07172360
Title: A Multicenter, Randomized, Double-blind, Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of VC005 Tablets in Subjects With Active Ankylosing Spondylitis
Brief Title: Efficacy and Safety Phase III Clinical Study of VC005 Tablets in Subjects With Active Ankylosing Spondylitis.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VC005-301
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Active Ankylosing Spondylitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VC005 Tablets Low Dose groups (Experimental)
  Interventions: Drug: VC005 tablets
- VC005 Tablets High Dose groups (Experimental)
  Interventions: Drug: VC005 tablets
- VC005 Tablets Placebo groups (Placebo Comparator)
  Interventions: Drug: VC005 Tablets Placebo

INTERVENTIONS:
Drug: VC005 tablets — VC005 groups repeat administration for 48 weeks
  Arms: VC005 Tablets High Dose groups; VC005 Tablets Low Dose groups
Drug: VC005 Tablets Placebo — VC005 placebo groups repeat administration for 48 weeks
  Arms: VC005 Tablets Placebo groups

SUMMARY:
This clinical trial is a multicenter, randomized, double-blind, controlled phase III clinical study.

ELIGIBILITY:
Inclusion Criteria:

* The subject understands and voluntarily signs the informed consent form (ICF) and is willing and able to comply with the study protocol;
* The subject is between 18 and 70 years of age (including borderline values) at the time of signing the ICF, regardless of gender;
* The subject has been diagnosed with AS according to the 1984 New York Revised Criteria for Ankylosing Spondylitis

Exclusion Criteria:

* Those who may be allergic to VC005, similar drugs or their excipients.
* Individuals who have undergone organ transplantation in the past and require continuous use of immunosuppressants.
* Those who, for any reason, are considered by the investigator to be unsuitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-12-26 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving an Assessment of disease activity (signs and symptoms) in ankylosing spondylitis 20% improvement (ASAS20) in response at week 12 of treatment. | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Principal Investigator — Peking University People's Hospital; Xu Liu, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China